CLINICAL TRIAL: NCT03323866
Title: Randomized Controled Double-blinded Study Comparing Mometasone Nasal Spray to Budesonide Irrigations in Patients With Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: Mometasone vs Budesonide in CRS With Polyposis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie Bussières, Otolaryngologist, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-1569
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Chronic Rhinosinusitis (Diagnosis), Nasal Polyposis
MeSH Terms: conditions — Disease; Nasal Polyps | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing mometasone nasal spray to budesonide irrigations for treatment of chronic rhinosinusitis with nasal polyposis
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mometasone nasal spray (Active Comparator): Mometasone nasal spray 50 mcg/dose, 2 sprays/nostril twice daily x 3 months Patients will also be taking Sinus Rinse once daily throughout the study period
  Interventions: Drug: Mometasone nasal spray
- Budesonide irrigation (Experimental): 2 cc budesonide nebule (0,5 mg/cc) incorporated to 240 of saline water (Sinus Rinse) to be taken on a daily basis x 3 months
  Interventions: Drug: Budesonide 0.5 MG/ML

INTERVENTIONS:
Drug: Budesonide 0.5 MG/ML — 2 cc nebule of budesonide in 240 cc of saline water (Sinus Rinse) once daily
  Arms: Budesonide irrigation
Drug: Mometasone nasal spray — Mometasone 50 mcg/spray 2 sprays twice daily
  Arms: Mometasone nasal spray

SUMMARY:
The principal objective is to compare the use of mometasone nasal spray to budesonide irrigations in patients suffering from CRSwNP who have never been operated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis with nasal polyps
* Absence of active infection at start of study

Exclusion Criteria:

* Diagnosis of chronic rhinosinusitis without nasal polyps
* Diagnosis of recurrent acute bacterial rhinosinusitis
* Previous sinus surgery (septal of inferior turbinate surgeries are not considered sinus surgeries)
* Cystic fibrosis or ciliary dyskinesia
* Allergy to corticosteroids
* Pregnant or lactating women
* Contra-indication to intranasal steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Disease specific quality of life questionnaire | 3 months after beginning of treatment
  SinoNasal Outcome Test - 22 This is a symptom score ranging from 0 to 110 points, 0 representing the absence of nasal symptoms and 110 being the most severe symptoms.

SECONDARY OUTCOMES:
Endoscopic evaluation of the nasal cavities | 3 months after beginning of treatment
  Lund Kennedy Endoscopic Score This is a score evaluating the healing of sinonasal cavities from 0 point (normal and healthy looking cavity) to 20 points (the most diseased cavity).

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada